CLINICAL TRIAL: NCT05266703
Title: Defining the Serum Ferritin Concentration in Kenyan Women at Which the Body Senses Iron Depletion and Begins to Upregulate Iron Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Jomo Kenyatta University of Agriculture and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PILLAR
Record Dates: First submitted 2022-02-08; First posted 2022-03-04 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Iron-deficiency; Ferritin Threshold; Iron Absorption; Stable Iron Isotopes
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Isotopically labelled iron sulfate 15mg (Other)
  Interventions: Other: Isotopically labelled iron sulfate 15mg

INTERVENTIONS:
Other: Isotopically labelled iron sulfate 15mg — test drink: water containing isotopic iron solution with vitamin C

SUMMARY:
The serum or plasma ferritin concentration (referred to hereafter as ferritin) is the most widely used indicator to detect iron deficiency and a low ferritin indicates depleted iron stores. However, the threshold ferritin that defines iron deficiency remains unclear and diagnostic ferritin cutoffs from expert groups vary widely.

Our study aim is to define the ferritin in Kenyan young women at which the body senses iron depletion and begins to upregulate iron absorption from the diet; this approach could provide a functionally defined threshold of iron deficiency in Sub-Saharan African women.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-28 y, not pregnant or lactating
* Body weight <75 kg
* body mass index (BMI) between 17 and 25 kg/m2
* No acute illness/infection (self-reported)
* No metabolic or gastrointestinal disorders (self-reported)
* No use of medications affecting iron absorption or metabolism during the study
* No intake of mineral/vitamin supplements 2 weeks prior to the first study visit and during the study

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption | Day 14
  shift in iron isotopic ratios measured in red blood cells

SECONDARY OUTCOMES:
Plasma Ferritin | Day 0
Plasma Ferritin | 4 months after isotope administration
Plasma Ferritin | 8 months after isotope administration
Plasma Ferritin | 12 months after isotope administration
soluble transferrin receptor | Day 0
soluble transferrin receptor | 4 months after isotope administration
soluble transferrin receptor | 8 months after isotope administration
soluble transferrin receptor | 12 months after isotope administration
C-reactive protein | Day 0
C-reactive protein | 4 months after isotope administration
C-reactive protein | 8 months after isotope administration
C-reactive protein | 12 months after isotope administration
alpha-1-glycoprotein | Day 0
alpha-1-glycoprotein | 4 months after isotope administration
alpha-1-glycoprotein | 8 months after isotope administration
alpha-1-glycoprotein | 12 months after isotope administration
Hemoglobin | Day 0
Hemoglobin | 4 months after isotope administration
Hemoglobin | 8 months after isotope administration
Hemoglobin | 12 months after isotope administration
Plasma Hepcidin | Day 0
Isotopic composition of red blood cells | 4 months after isotope administration
  shift in iron isotopic ratios measured in red blood cells
Isotopic composition of red blood cells | 8 months after isotope administration
  shift in iron isotopic ratios measured in red blood cells
Isotopic composition of red blood cells | 12 months after isotope administration
  shift in iron isotopic ratios measured in red blood cells

CONTACTS AND LOCATIONS:
Locations (1):
- Msambweni County Referral Hospital, Msambweni, Kenya

IPD SHARING:
Plan to Share IPD: No